CLINICAL TRIAL: NCT04719910
Title: The Putative Role of the Pavlovian Reflex as a Non-pharmacological Preoperative Intervention in the Prevention of Postoperative Nausea and Vomiting
Brief Title: Food Related Video and the Incidence of Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ANES-2021-29548
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The study group will watch 15 minute long videos of cooking and preparing the food of the patient's preferred type of food prior to be taken to the operating room.
  Interventions: Other: Visual exposure to taped food preparation
- Placebo group (Placebo Comparator): The control group will watch 15 minute long non-food related videos.
  Interventions: Other: Visual exposure to topics not related to food

INTERVENTIONS:
Other: Visual exposure to taped food preparation — Patients in the study group can watch the preparation of the the type of food she prefers to eat normally.
  Arms: Study group
Other: Visual exposure to topics not related to food — Patients in the placebo group can choose a video that is relaxing but not related to food.
  Arms: Placebo group

SUMMARY:
Postoperative nausea/vomiting (PONV) is a common problem following surgery and anesthesia. There are risk factors that increase the incidence of PONV that are related to the patient, to the surgical procedure or to the anesthetic agents. At the subjective level PONV is described as worse and more feared than postoperative pain by many patients. At the objective level it increases the length of stay in the recovery room, it results in unplanned hospital admission and Emergency Room visits, and therefore increased cost of care. A lot of research work has been done to identify pharmacological agents to prevent and treat PONV. The higher the risk of a patient the higher number of these drugs are combined for prophylaxis. However, these drugs have significant side effects of their own. Much less attention has been paid to potential non-pharmacological PONV prevention options. The purpose of our study is to investigate the putative role of the natural stimulation of normal gastrointestinal function via the Pavlovian reflex. We seek to find a natural method with no side effects to improve PONV prophylaxis in patients with risk factors for that postoperative complication.

DETAILED DESCRIPTION:
The study will be conducted in 18-40 years old female volunteers who are undergoing planned, elective, non-cancer surgical procedure as outpatients, and who are identified to have either history or significant risk of PONV. The latter will be calculated by the questionnaire we currently use during our routine preoperative anesthesia evaluation (see in detail below in the Study design section).

Patients who meet the study enrollment criteria will be identified on the surgical schedule the day before the planned intervention. The recruitment will occur during the preoperative admission process.

These patients will be randomly assigned to either the study group or to the control group. The study group will watch videos of preparation and cooking of their favorite foods while waiting for their surgery. Patients in the control group will watch videos that are not food related.

The anesthesia team in the OR and the PACU team who manages the patient's postoperative recovery will be blinded to which group the patient is enrolled to. The intraoperative antiemetics will be provided by the study team as outlined in the Study design section below.

The anesthesia protocol will be standardized. All patient who are enrolled in the study will require general anesthesia with endotracheal intubation. After intravenous induction, muscle relaxation with rocuronium and intubation of the trachea anesthesia will be maintained with sevoflurane and opioid boluses for analgesia as deemed necessary by the anesthesia team. Antiemetics (as described below) will be administered 30 minutes prior to planned emergence, residual muscle relaxant will be reversed with sugammadex.

The patients will be taken to the recovery room. Beyond their routine vital sign and pain score monitoring and observation the occurrence and degree of nausea and vomiting, as well as the time to discharge to home or unplanned admission due to therapy resistant vomiting will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old female
* American Society of Anesthesiologists Physical Status I and II
* Personal history of postoperative nausea and vomiting
* Personal history of motion sickness
* Non-smoker status
* Undergoing scheduled elective surgical procedures and general anesthesia for non-cancer surgery of:
* breast
* gynecology
* ear, nose and throat
* eye
* Duration of surgery less than 3 hours will be enrolled in the study.

Exclusion Criteria:

* Ages older than 40 years and younger than 18 years
* Morbid obesity (BMI > 35 kg/m2)
* Uncontrolled gastroesophageal reflux disease (GERD)
* Smoking
* Cancer and chemotherapy
* Vertigo
* Meniere's disease
* Pseudotumor cerebri and other central nervous diseases that may induce nausea and vomiting
* Prolonged (> 15 minutes) intraoperative hypotension
* Estimated blood loss > 20 % of estimated blood volume
* Emergency surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Change of the incidence of postoperative vomiting | Immediately postoperative
  The number of the episodes of emesis will be counted and recorded in the patients' records.
Change of postoperative anti emetic drug administration | Immediate postoperative
  The type and dose of administered antiemetic drugs will be recorded and analyzed in the patients' charts.

SECONDARY OUTCOMES:
Change of recovery room length of stay | Immediate postoperative
  The time between arriving to and discharge from the recovery room will be recorded in the patients' charts.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amirshahi M, Behnamfar N, Badakhsh M, Rafiemanesh H, Keikhaie KR, Sheyback M, Sari M. Prevalence of postoperative nausea and vomiting: A systematic review and meta-analysis. Saudi J Anaesth. 2020 Jan-Mar;14(1):48-56. doi: 10.4103/sja.SJA_401_19. Epub 2020 Jan 6. PMID 31998020
- [Background] Hirsch J. Impact of postoperative nausea and vomiting in the surgical setting. Anaesthesia. 1994 Jan;49 Suppl:30-3. doi: 10.1111/j.1365-2044.1994.tb03580.x. PMID 8129160
- [Background] Macario A, Weinger M, Carney S, Kim A. Which clinical anesthesia outcomes are important to avoid? The perspective of patients. Anesth Analg. 1999 Sep;89(3):652-8. doi: 10.1097/00000539-199909000-00022. PMID 10475299
- [Background] Habib AS, Chen YT, Taguchi A, Hu XH, Gan TJ. Postoperative nausea and vomiting following inpatient surgeries in a teaching hospital: a retrospective database analysis. Curr Med Res Opin. 2006 Jun;22(6):1093-9. doi: 10.1185/030079906X104830. PMID 16846542
- [Background] Fortier J, Chung F, Su J. Unanticipated admission after ambulatory surgery--a prospective study. Can J Anaesth. 1998 Jul;45(7):612-9. doi: 10.1007/BF03012088. PMID 9717590
- [Background] Dzwonczyk R, Weaver TE, Puente EG, Bergese SD. Postoperative nausea and vomiting prophylaxis from an economic point of view. Am J Ther. 2012 Jan;19(1):11-5. doi: 10.1097/MJT.0b013e3181e7a512. PMID 20634672
- [Background] Apfel CC, Korttila K, Abdalla M, Kerger H, Turan A, Vedder I, Zernak C, Danner K, Jokela R, Pocock SJ, Trenkler S, Kredel M, Biedler A, Sessler DI, Roewer N; IMPACT Investigators. A factorial trial of six interventions for the prevention of postoperative nausea and vomiting. N Engl J Med. 2004 Jun 10;350(24):2441-51. doi: 10.1056/NEJMoa032196. PMID 15190136
- [Background] Gan TJ. Mechanisms underlying postoperative nausea and vomiting and neurotransmitter receptor antagonist-based pharmacotherapy. CNS Drugs. 2007;21(10):813-33. doi: 10.2165/00023210-200721100-00003. PMID 17850171
- [Background] Lee A, Done ML. The use of nonpharmacologic techniques to prevent postoperative nausea and vomiting: a meta-analysis. Anesth Analg. 1999 Jun;88(6):1362-9. doi: 10.1097/00000539-199906000-00031. PMID 10357346
- [Background] Darvall JN, Handscombe M, Leslie K. Chewing gum for the treatment of postoperative nausea and vomiting: a pilot randomized controlled trial. Br J Anaesth. 2017 Jan;118(1):83-89. doi: 10.1093/bja/aew375. PMID 28039245
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Pierre S, Benais H, Pouymayou J. Apfel's simplified score may favourably predict the risk of postoperative nausea and vomiting. Can J Anaesth. 2002 Mar;49(3):237-42. doi: 10.1007/BF03020521. PMID 11861340
- [Background] Sherif L, Hegde R, Mariswami M, Ollapally A. Validation of the Apfel Scoring System for Identification of High-risk Patients for PONV. Karnataka Anaesth J. 2015;1(3):115-117
- [Background] Davis CJ, Lake-Bakaar GV, Grahame-Smith DG. Nausea and Vomiting: Mechanisms and Treatment. Springer Science & Business Media; 2012
- [Background] Stern RM, Jokerst MD, Levine ME, Koch KL. The stomach's response to unappetizing food: cephalic-vagal effects on gastric myoelectric activity. Neurogastroenterol Motil. 2001 Apr;13(2):151-4. doi: 10.1046/j.1365-2982.2001.00250.x. PMID 11298993
- [Background] Sarles H, Dani R, Prezelin G, Souville C, Figarella C. Cephalic phase of pancreatic secretion in man. Gut. 1968 Apr;9(2):214-21. doi: 10.1136/gut.9.2.214. No abstract available. PMID 5655031